CLINICAL TRIAL: NCT07161336
Title: Role of Methotrexate in Ultrasound Proven Synovitis in Patients With Knee Osteoarthritis : A Randomized Controlled Trial
Brief Title: Role of Methotrexate in Ultrasound Proven Synovitis in Primary Knee OA
Acronym: MTX in knee OA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Akash Ahmed Alif, MD resident , Rheumatology department, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5535
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Osteo Arthritis of the Knee; Synovitis of Knee; Methotrexate
Keywords: knee OA; synovitis; Methotrexate
MeSH Terms: conditions — Synovitis | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: A Double blind randomized controlled trial study will be carried out in the outpatient department of rheumatology in BMU to determine the efficacy of Methotrexate in the treatment of primary knee OA associated with synovitis. Ethical approval will be taken from the Ethical Review Committee of BMU, Dhaka. At first, patients who attend the outpatient rheumatology department with knee pain will be requested to give verbal consent. Then, primary knee OA will be diagnosed by ACR clinical and radiological criteria, and subsequently, history, physical examination, and investigation will be done for evaluation of exclusion criteria. Then MSKUS examinations of knee joint and scoring (OMERACT SCORE) will be performed to detect synovitis by one rheumatologist experienced in MSK ultrasound using a MINDRAY machine with an 6-18 MHz linear array transducer operating at 3 MHz Power Doppler (PD) signal settings will be Pulse repetition frequency 750Hz, Doppler frequency 11.1 MHz, gain of 50% and low wa
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methotrexate (MTX) (Active Comparator): As it will be a double blinded study , the investigator and the patient is unable to know if the drug is MTX or placebo
  Interventions: Drug: Methotrexate (MTX)
- Placebo (Placebo Comparator): As it will be a double blinded study , the investigator and the patient is unable to know if the drug is MTX or placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate (MTX) — One group will receive MTX, starting with 15 mg per week for the first 2 weeks then increase to 20 mg and continue for the remaining period if tolerated. another group will receive placebo
  Other Names: MTX; Low dose Methotrexate
  Arms: Methotrexate (MTX)
Drug: Placebo — The investigational drug and the placebo will be formulated to be identical in appearance, packaging, labeling. Blinded study medications will be prepared, packaged, and labeled by the sponsor according to Good Manufacturing Practice (GMP) standards. All packaging will use neutral labeling with unique subject numbers only.
  Arms: Placebo

SUMMARY:
Background:

Osteoarthritis (OA) is a leading cause of disability worldwide, with limited treatment options and many patients suffering from chronic pain. Modern imaging has revealed that OA involves complex changes in cartilage, subchondral bone, and synovium. Pain in OA is often linked to synovitis, which is common in the condition. Methotrexate (MTX), a proven treatment for synovitis in inflammatory arthritis like rheumatoid arthritis and has a well-known safety profile. The proposal suggests that using MTX may have potential to treat symptomatic knee OA with USG (musculoskeletal ultrasound) proven synovitis by reducing synovitis and as a result, alleviate pain.

Objectives:

To assess the role of methotrexate in primary knee osteoarthritis associated with ultrasound proven synovitis.

Methods:

This randomized Controlled trial will be conducted in the department of Rheumatology, Bangladesh Medical University (BMU) from July 2025 to June 2026. A total of 70 patients will be enrolled with primary knee OA diagnosed on the basis of ACR Criteria for Knee OA with informed written consent. MSK USG examinations of knee joint and scoring (OMERACT SCORE) will be performed to detect synovitis by a rheumatologist expert in MSK US. Then randomization will be done into group A and group B following a randomization table, each consisting of 35 patients. Consecutive sampling techniques will be followed. One group will receive MTX (start with 15 mg per week for the first 2 weeks then increase to 20 mg and continue for the remaining period if tolerated) and Both groups of patients will be allowed to take NSAIDs on a requirement basis with documentation and follow non-pharmacological treatment of OA. At the end of 3rd and 6th month pain and functional status will be assessed by WOMAC, VAS and quality of life will be assessed by using Bangla version of SF-12. At the end of 6th month improvement of synovitis will be seen by MSK USG of involved knees with OMERACT scoring. Primary endpoint for efficacy will be assessed at the end of 24th week by WOMAC. Secondary endpoints will be determined by VAS and SF-12. Adverse effects will be assessed by history, physical examinations and investigations. The data will be analyzed by using the latest version SPSS software (Version 29). Results will be recorded using means and standard deviations. Results will be compared among two groups with a 95% confidence interval and a p- value of < 0.05 will be considered statistically significant. The degrees of statistical significance between groups will be analyzed by unpaired t test (for quantitative normally distributed data) and Mann Whitney U test if there is skewed distribution. Qualitative data in between groups will be analyzed by the chi square test. Probabilities of associations will be assessed by calculating Pearson's rank correlation coefficient. P-value <0.05 will be regarded as statistically significant. The nature, purpose and implication of the study as well as the entire spectrum of benefits and risks of study will be explained to the patients. Privacy and confidentiality of the subject will be maintained. Each patient will enjoy the right to participate and or withdraw from the study at any point of the study period. Ethical clearance will be obtained from the institutional Review Board (IRB) of BMU.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 40 to 70 years
* Patients fulfilling American College of Rheumatology (ACR) clinical and radiological criteria for knee OA. (knee pain + at least 3 of 5 that not including "no palpable warmth")
* Knee pain on most days for at least 6 months, with a pain VAS of at least 40mm
* Radiological grading of OA with Kallgren-Lawrence grade of 2 to 3
* Patients with the presence of knee synovitis in Musculoskeletal ultrasound

Exclusion Criteria:

* Any known inflammatory arthritis
* BMI >= 40 kg/m2
* Abnormal renal (e.g. abnormal renal function Creatinine clearance <35 ml) hepatic (including active hepatitis B, hepatitis C, abnormal liver function), hematological (e.g. white cell count < 4 × 109/L, platelets <100 ×109/L, or hemoglobin < 9 g/dL), function
* Use of intra-articular, intramuscular or oral corticosteroids in previous 4 weeks
* History knee joint surgery, Charcot joint
* Severe valgus knee deformity (angle of genu valgum > 30°)
* Use of any disease modifying agents (e.g. hydroxychloroquine or sulfasalazine) in previous 3 months
* Allergic to MTX
* Pregnant or lactating women

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
To assess the role of Methotrexate to change the functional status with Western Ontario and McMaster Universities Osteoarthritis Index in patients with ultrasound proven synovitis associated with primary knee Osteoarthritis. | 6 months
  This Western Ontario and McMaster Universities Osteoarthritis Index have 24 questions divided in 3 domains ( PAIN, Stiffness, Difficulty in performing daily activities) each of the 24 questions having a visual analog scale of 0-10.Patients will score themselves between 0-10 for each question . So the minimum score will be 0 and the maximum score will be 240 .The higher the number more severe the condition.

SECONDARY OUTCOMES:
changes in synovitis by Outcome Measures in Rheumatology (OMERACT) scoring in patients with primary knee OA. | 6 months
  Outcome Measures in Rheumatology (OMERACT) scoring of USG findings of knee joint have 7 domains , each of the domains will be scored based on the ultrasound findings like the following.
  USG findings
  1. Synovitis 0 1 2 3
  2. Cartilage damage 0 1 2 3
  3. Meniscal damage 0 1 2
  4. Osteophytes : 0 1 2 3
  5. Synovial hypertrophy : Present=1or Absent=0
  6. Effusion : Present=1 or Absent=0
  7. Synovial PD signal : Present=1 or Absent=0
  The higher the number more severe the condition
Change in Quality of life through 12-item Short-Form Health Survey (SF-12) in patients with primary knee OA | 6 months
  The 12-Item Short Form Survey (SF-12v2) is a 12- item questionnaire used to assess generic health outcomes from a patient's perspective. SF-12 is used to measure physical and mental components of health in patients with any chronic illness on a broad range of functional domains. The SF-12 consists of a subset of 12 items drawn from SF-36. covering the same eight domains of health outcomes measuring physical functioning (PF), role physical (RP, physical health problems), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE, emotional problems) and mental health (MH). Higher scores represent better health status. Score more than 50 is better and below 50 is considered lower than average.

CONTACTS AND LOCATIONS:
Overall Officials: Shamim Ahmed Professor, FCPS, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh, Dhaka, Dhaka Division, Bangladesh